CLINICAL TRIAL: NCT03635398
Title: Intranasal Midazolam for Pediatric Pre-procedural Sedation and Pre-procedural Anti-anxiety Using sipNose Device - a Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: SipNose (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RMC-17-0435
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Procedural Sedation; Intra-nasal Delevery Device
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intranasal Midazolam by SipNose device (Experimental)
  Interventions: Device: Sipnose device
- Intranasal Midazolam by MAD (Mucosal Atomization Device) (Active Comparator)
  Interventions: Device: MAD (Mucosal Atomization Device)
- oral administration of midazolam (Active Comparator)
  Interventions: Drug: midazolam

INTERVENTIONS:
Device: Sipnose device — SipNose's intranasal drug delivery platform uses an innovative mechanism that is suposed to improves efficacy, patient compliance and safety
  Arms: Intranasal Midazolam by SipNose device
Device: MAD (Mucosal Atomization Device) — MAD (Mucosal Atomization Device)
  Arms: Intranasal Midazolam by MAD (Mucosal Atomization Device)
Drug: midazolam — oral administration of midazolam
  Arms: oral administration of midazolam

SUMMARY:
A Three-arm, Randomized Controlled Trial for Pediatric Pre-procedural Sedation and Pre-procedural Anti-anxiety: Intranasal Midazolam by SipNose versus MAD Versus oral administration

ELIGIBILITY:
Inclusion Criteria:

* every child >1y who is intended for medical procedure in the emrgency room(suce as: IV insertion, blood sample collection, urinary catether insertion, laceration repair

Exclusion Criteria:

* ASA>2
* Active respiratory infection
* systemic illness
* Allergy to Midazolam

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Anexiety level | within 60 minute
  measured by modified PREOPERATIVE ANXIETY SCALE (YALE)
Sedation level | within 60 minute
  measured by RAMSAY SEDATION SCALE

CONTACTS AND LOCATIONS:
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No
Because of commercial confidentially the study database will not become public within the first 3 years since the begining of the study